CLINICAL TRIAL: NCT01336634
Title: A Phase II Study of the BRAF Inhibitor Dabrafenib as a Single Agent and in Combination With the MEK Inhibitor Trametinib in Subjects With BRAF V600E Mutation Positive Metastatic (Stage IV) Non-small Cell Lung Cancer
Brief Title: Study of Selective BRAF Kinase Inhibitor Dabrafenib Monotherapy Twice Daily and in Combination With Dabrafenib Twice Daily and Trametinib Once Daily in Combination Therapy in Subjects With BRAF V600E Mutation Positive Metastatic (Stage IV) Non-small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113928; 2011-001161-41 (EudraCT Number); CDRB436E2201 (Other: Novartis)
Record Dates: First submitted 2011-04-07; First posted 2011-04-18 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: BRAF V600E; trametinib; dabrafenib; GSK2118436; GSK1120212; Oncology; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Dabrafenib Monotherapy) (Experimental): Participants received Dabrafenib 150mg BID and continued treatment until disease progression, death, or unacceptable adverse event.
  Participants receiving and adequately tolerating dabrafenib as a single agent and who continue to meet the inclusion and exclusion criteria had the option to switch to Dabrafenib (150 mg BID) and Trametinib (2 mg once daily) combination treatment within 4 weeks of radiologic disease progression with prior approval from a medical monitor.
  Interventions: Drug: Dabrafenib
- Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E (Experimental): Participants received Dabrafenib 150 mg BID in combination with Trametinib 2 mg once daily and continued treatment until disease progression, death, or unacceptable adverse event.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Cohort C - Double Combination (Dabrafenib+Trametinib) naive mBRAF V600E (Experimental): Participants received Dabrafenib 150 mg BID in combination with Trametinib 2 mg once daily and continued treatment until disease progression, death, or unacceptable adverse event.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib study treatment was provided as 50 mg and 75 mg hydroxypropyl methylcellulose (HPMC) capsules. Each capsule contains 50 mg or 75 mg of free base (present as the mesylate salt)
  Other Names: DRB436; GSK2118436
Drug: Trametinib — Trametinib study treatment was provided as 0.5 mg and 2 mg tablets. Each tablet contained 0.5 mg or 2 mg of trametinib parent (present as the dimethyl sulfoxide solvate)
  Other Names: TMT212; GSK1120212
  Arms: Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E; Cohort C - Double Combination (Dabrafenib+Trametinib) naive mBRAF V600E

SUMMARY:
This was a Phase II, multicenter, non-randomized, open-label study to assess the efficacy, safety, and tolerability of dabrafenib administered as a single agent and in combination with trametinib in stage IV disease to subjects with BRAF mutant advanced non-small cell lung cancer. Central confirmation testing for the BRAF V600E mutation was performed and a sufficient number of subjects were enrolled with the intent of having at least 125 centrally confirmed subjects among the three cohorts.

DETAILED DESCRIPTION:
Subjects enrolled in Cohort A (Monotherapy Population) were required to have relapsed or progressed on at least one platinum based chemotherapy regimen prior to enrollment (i.e. dabrafenib was no less than second line treatment for metastatic disease). Additional lines of prior anti-cancer therapy were allowed. Subjects received dabrafenib as a single agent at the recommended dose of 150 mg twice daily. A 2 stage design with a planned sample size of 40 subjects was initially used for Cohort A.

Subjects enrolled in Cohort B (Combination Second-Line Population) were required to have relapsed or progressed on at least one platinum based chemotherapy prior to enrollment but did not receive more than 3 prior systemic anti-cancer therapies (i.e. dabrafenib/trametinib were second, third, or fourth line treatment for metastatic disease). Subjects received the recommended dose of both drugs (dabrafenib 150 mg twice daily and trametinib 2 mg once daily).

Subjects enrolled in Cohort C (Combination First-Line Population) did not receive prior systemic anti-cancer therapies for metastatic disease (i.e. dabrafenib/trametinib was first line treatment for metastatic disease). Subjects received the recommended dose of both drugs (dabrafenib 150 mg twice daily and trametinib 2 mg once daily).

Crossover: Subjects receiving and adequately tolerating dabrafenib as a single agent and who continued to meet the inclusion and exclusion criteria (including the additional criteria for combination therapy) had the option to crossover to dabrafenib (150 mg BID) and trametinib (2 mg once daily) combination treatment at the time of radiologic disease progression with prior approval from a Medical Lead. If a subject was receiving less than 150 mg BID of dabrafenib at the time of the crossover, the subject was to continue at the lower dose of dabrafenib when initiating combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Histologically or cytologically confirmed non-small cell cancer of the lung (NSCLC) stage IV (accordingto AJCC Staging 7th Edition);
* For Cohorts A and B, documented tumor progression (based on radiological imaging) after receiving at least one prior approved platinum-based chemotherapy regimen for advanced stage/metastatic NSCLC. An alternate chemotherapeutic agent/regimen is an acceptable substitute in the event that the subject was intolerant to, or ineligible to receive platinum based chemotherapy. Subjects enrolled in Cohort B cannot have more than 3 prior systemic treatments for advanced stage/metastatic NSCLC (neoadjuvant and adjuvant therapies are not counted in number of prior regimens and maintenance therapy is not counted as a separate regimen). Subjects in Cohort C will be required to have not received prior systemic anti-cancer therapies for metastatic disease (i.e., dabrafenib/trametinib will be 1st line treatment for metastatic disease);
* Measurable disease according to Response Evaluation Criteria in Solid Tumors [RECIST 1.1];
* At least 18 years of age;
* Anticipated life expectancy of at least three months;
* Presence of a BRAF V600E mutation in lung cancer tissue. Mutation must be locally confirmed in a CLIA-certified laboratory (or equivalent). An adequate amount of tumor tissue (archived tumor tissue, or fresh biopsy if archived tissue is not available) must be available at the time of enrolment for central validation of BRAF mutation;
* Able to swallow and retain oral medication;
* Women of childbearing potential must have a negative serum pregnancy test within 14 days before the first dose of study treatment and agree to use effective contraception during the study; NOTE: Oral contraceptives are not reliable due to potential drug-drug interaction with dabrafenib.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2;
* Must have adequate organ function as defined by the following baseline values:

Absolute neutrophil count (ANC) >/=1.5x10^9/L Hemoglobin >/=9 g/dL Platelets >/=100x10^9/L Prothrombin time /International normalized ratio (INR) and partial thromboplastin time </=1.5xULN (Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to starting study treatment.) Total bilirubin </=1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5xULN Serum creatinine </=1.5 mg/dL (if serum creatinine is >1.5 mg/dL, calculate creatinine clearance using standard Cockcroft and Gault; creatinine clearance must be > 50 mL/min); creatinine clearance should be >/= 50 mL/min Left ventricular ejection fraction >/= institutional lower limit of normal ECHO

* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category
* Previously tested for presence of EGFR and ALK mutations in lung cancer tissue confirmed in a CLIA-certified laboratory (or equivalent). Subjects with EGFR or ALK mutation are eligible if they have previously received EGFR or ALK inhibitor(s) respectively.

Exclusion Criteria:

* Previous treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, LGX818, and XL281/BMS-908662) or MEK inhibitor (including but not limited to trametinib, AZD6244, and RDEA119) prior to start of study treatment (Note: Prior treatment with dabrafenib is allowed for crossover subjects in Cohort A);
* Anti-Cancer therapy including chemotherapy, radiation-therapy, immunotherapy, biologic therapy or major surgery within 14 days prior to start of study treatment (Note: Dabrafenib monotherapy within 14 days prior to starting combination therapy is allowed for crossover subjects in Cohort A);
* Use of any investigational anti-cancer drug within 14 days or 5-half-lives (minimum 14 days), prior to start of study medication (Note: Dabrafenib monotherapy within 14 days prior to starting combination therapy is allowed for crossover subjects in Cohort A);
* Current use of a prohibited medication or expected to require any of these medications during treatment with study treatment.
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) Grade 2 or higher from previous anti-cancer therapy, except alopecia;
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK medical monitor for guidance to enrol the subject;
* Known Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection. Subjects with laboratory evidence of cleared HBV and HCV infection may be enrolled;
* History of another malignancy < 3 years prior to starting study treatment or any malignancy with confirmed activating RAS-mutation; Exceptions: Subjects with any of the following malignancies within 3 years (does not include malignancies with confirmed activating RAS-mutation) are eligible: (a) a history of completely resected skin cancer, (b) successfully treated in situ carcinoma, (c) chronic lymphocytic lymphoma (CLL) in stable remission, or (d) indolent prostate cancer (definition: clinical stage T1 or T2a, Gleason score <= 6, and prostate specific antigen [PSA] < 10 ng/mL) requiring no or only anti-hormonal therapy with histologically confirmed tumour lesions that can be clearly differentiated from lung cancer target and non-target lesions are eligible
* Subjects with brain metastases are excluded if their brain metastases are:
* Symptomatic OR
* Treated (surgery, radiation therapy) but not clinically and radiographically stable 3 weeks after local therapy(as assessed by contrast enhanced magnetic resonance imaging [MRI] or computed tomography [CT]), OR
* Asymptomatic and untreated but >1 cm in the longest dimension
* A history or evidence of cardiovascular risk including any of the following:

Corrected QT (QTc) interval >=480 msecs History of acute coronary syndromes (including myocardial infarction or unstable angina) within 6 months prior to first dose of study treatment Coronary angioplasty, or stenting within the past 24 weeks; A history or evidence of current Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) guidelines; Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic >90 mmHg which cannot be controlled by antihypertensive therapy; Abnormal cardiac valve morphology ( >=Grade 2) documented by echocardiogram (subjects with Grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study; Patients with intra-cardiac defibrillators A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Subjects with atrial fibrillation controlled for > 30 days prior to randomization are eligible.

Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension, etc.), psychological, familial, sociological, or geographical conditions that interfere with the subject's safety or obtaining informed consent or do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol;

* Pregnant, or actively breastfeeding females.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Additional Exclusion Criteria for dabrafenib and trametinib combination therapy (Cohort B and C as well as subjects that crossover from monotherapy to combination therapy):
* History of interstitial lung disease or pneumonitis
* A history or current evidence of retinal vein occlusion (RVO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-08-05 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- United States (14):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- France (8):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Moers
- Italy (2):
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Orbassano
- Japan (2):
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Seoul, South Korea
- Spain (5):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Seville
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Schadendorf D, Robert C, Dummer R, Flaherty KT, Tawbi HA, Menzies AM, Banerjee H, Lau M, Long GV. Pyrexia in patients treated with dabrafenib plus trametinib across clinical trials in BRAF-mutant cancers. Eur J Cancer. 2021 Aug;153:234-241. doi: 10.1016/j.ejca.2021.05.005. Epub 2021 Jul 2. PMID 34225229
- [Derived] Li J, Sasane M, Zhang J, Zhao J, Ricculli ML, Yao Z, Redhu S, Signorovitch J. Is time to progression associated with post-progression survival in previously treated metastatic non-small cell lung cancer with BRAF V600E mutation? A secondary analysis of phase II clinical trial data. BMJ Open. 2018 Aug 17;8(8):e021642. doi: 10.1136/bmjopen-2018-021642. PMID 30121602
- [Derived] Planchard D, Smit EF, Groen HJM, Mazieres J, Besse B, Helland A, Giannone V, D'Amelio AM Jr, Zhang P, Mookerjee B, Johnson BE. Dabrafenib plus trametinib in patients with previously untreated BRAFV600E-mutant metastatic non-small-cell lung cancer: an open-label, phase 2 trial. Lancet Oncol. 2017 Oct;18(10):1307-1316. doi: 10.1016/S1470-2045(17)30679-4. Epub 2017 Sep 11. PMID 28919011
- [Derived] Planchard D, Besse B, Groen HJM, Souquet PJ, Quoix E, Baik CS, Barlesi F, Kim TM, Mazieres J, Novello S, Rigas JR, Upalawanna A, D'Amelio AM Jr, Zhang P, Mookerjee B, Johnson BE. Dabrafenib plus trametinib in patients with previously treated BRAF(V600E)-mutant metastatic non-small cell lung cancer: an open-label, multicentre phase 2 trial. Lancet Oncol. 2016 Jul;17(7):984-993. doi: 10.1016/S1470-2045(16)30146-2. Epub 2016 Jun 6. PMID 27283860
- [Derived] Planchard D, Kim TM, Mazieres J, Quoix E, Riely G, Barlesi F, Souquet PJ, Smit EF, Groen HJ, Kelly RJ, Cho BC, Socinski MA, Pandite L, Nase C, Ma B, D'Amelio A Jr, Mookerjee B, Curtis CM Jr, Johnson BE. Dabrafenib in patients with BRAF(V600E)-positive advanced non-small-cell lung cancer: a single-arm, multicentre, open-label, phase 2 trial. Lancet Oncol. 2016 May;17(5):642-50. doi: 10.1016/S1470-2045(16)00077-2. Epub 2016 Apr 11. PMID 27080216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 50 sites across 11 countries: Netherlands(2), United States(15), Germany(4), Spain(7), France(8), Italy(3), Taiwan(2), South Korea(3), United Kingdom(3), Japan(2), Norway(1)
Groups:
- Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID: Participants with or without prior systemic anti-cancer therapy received Dabrafenib 150 mg BID until disease progression, death, or unacceptable adverse event(s) (AEs) or investigator discretion to discontinue or decision to crossover from monotherapy to combination therapy.
- Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD: Participants who had received 1-3 prior lines of systemic anti-cancer therapies for advanced stage/metastatic disease received Dabrafenib 150 mg BID and Trametinib 2 mg once daily (OD). Treatment continued until disease progression, death, or unacceptable AEs or investigator discretion to discontinue.
- Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD: Participants who had not received any prior systemic anti-cancer for metastatic disease therapies were given Dabrafenib 150 mg BID and Trametinib 2 mg OD. Treatment continued until disease progression, death, or unacceptable AEs or at investigator discretion to discontinue.
Period: Overall Study
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Started (All participants who received at least one dose of study treatment were included in the All Treated Population (ATP)) | 84 | 57 | 36 (includes 34 subjects from Cohort C and 2 subjects enrolled as protocol deviations from Cohort B.)
2nd Line Plus All Treated (All Treated Population who had relapsed or progressed after receiving at least one line of prior anti-cancer therapy for metastatic disease.) | 78 | 57 | 0
1st Line All Treated (All Treated Population who had not received any prior anti-cancer therapy for metastatic disease.) | 6 | 2 | 34
Crossover (All Treated Population who were assigned to monotherapy cohort and elected to crossover to combination treatment following disease progression on monotherapy.) | 20 | 0 | 0
Completed (Study ended when progression of disease had occurred in all patients in Cohorts B and C, a minimum of 70% of subjects had died in each cohort, or five years had passed since the last subject's first dose, whichever came first.) | 70 | 49 | 27
Not Completed | 14 | 8 | 9
Not completed — Study closed/terminated | 5 | 6 | 6
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Total
Number analyzed (Participants) | 84 | 57 | 36 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (10.51) | 65.1 (10.14) | 67.8 (11.00) | 65.5 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 28 | 22 | 94
  Male | 40 | 29 | 14 | 83
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 64 | 49 | 30 | 143
  Asian | 18 | 4 | 3 | 25
  African American Heritage | 2 | 0 | 0 | 2
  Native Hawaiian or other Pacific islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 2 | 1 | 3
  Other | 0 | 2 | 1 | 3
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classifies participants according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). ECOG PS: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours
  Participants
    Grade 0 | 20 | 17 | 13 | 50
    Grade 1 | 52 | 35 | 22 | 109
    Grade 2 | 12 | 5 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR) by investigator assessment as per RECIST v1 .1 criteria. Specifically, ORR = (number of subjects with a confirmed best overall response of CR or PR) divided by the total number of subjects in the corresponding analysis population.
Time Frame: From study treatment start date until first documented complete response or partial response, assessed up to approximately 50 months
Population: All Treated Population (ATP).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A (Dabrafenib Monotherapy): Participants who have relapsed or progressed after receiving at least one line of prior anti-cancer therapy for metastatic disease received dabrafenib 150 mg BID. It was continued until disease progression or death or unacceptable AEs or investigator discretion to discontinue or decision to crossover from monotherapy to combination therapy.
- Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD: Crossover - Double Combination (Dabrafenib+Trametinib): Participants received Dabrafenib 150 mg BID in combination with Trametinib 2 mg once daily and continued treatment until disease progression, death, or unacceptable adverse event.
Arm/Group | Cohort A (Dabrafenib Monotherapy) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 78 | 57 | 36 | 20
Participants | 27 | 39 | 23 | 4

2. Secondary Outcome: Progression Free Survival (PFS) Based on Local Investigator Assessment
Description: Progression Free Survival (PFS) was defined as the time from study treatment start date to the date of first radiologically documented progression or death due to any cause. If a patient did not progress or die at the time of the analysis data cut-off or start of new antineoplastic therapy, PFS was censored at the date of the last adequate tumor assessment before the earliest of the cut-off date or the start date of additional anti-neoplastic therapy. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria RECIST v1.1, as 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline and/or unequivocal progression of the non-target lesions and/or appearance of a new lesion. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm.
Time Frame: From study treatment start date until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 113 months
Population: All Treated Population (ATP). Only participants with an evaluable PFS events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Dabrafenib Monotherapy) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 65 | 48 | 28 | 18
Months | 5.4 [2.8 to 6.9] | 10.2 [6.9 to 16.7] | 10.8 [7.0 to 14.5] | 11.0 [3.0 to 18.7]

3. Secondary Outcome: Duration of Response (DoR) Based on Local Investigator Assessment
Description: Duration of Response (DoR) was defined as the time from the first documented occurrence of response (PR or CR) until the date of the first documented progression based on RECIST v1.1 or death.
Time Frame: From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to approximately 113 months
Population: All Treated Population (ATP). Only responders (PR or CR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Dabrafenib Monotherapy) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 27 | 39 | 23 | 4
Months | 11.8 [5.4 to 23.5] | 9.8 [6.9 to 18.3] | 10.2 [8.3 to 15.2] | 13.4 [7.6 to 19.3]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from first dose until death due to any cause. If a patient was not known to have died at the time of analysis cut-off, OS was censored at the date of last contact.
Time Frame: From study treatment start date until date of of death from any cause, assessed up to approximately 113 months
Population: All Treated Population (ATP). No separate OS analysis was conducted for cross over patient, as they were included in Cohort A (Dabrafenib Monotherapy Second-Line Plus).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A (Dabrafenib Monotherapy) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 67 | 49 | 27
Months | 12.7 [7.3 to 16.3] | 18.2 [14.3 to 28.6] | 17.3 [12.3 to 40.2]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The distribution of adverse events (AE) was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 30 days safety follow-up, assessed up to approximately 81 months
Population: All Treated Population (ATP)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 84 | 57 | 36 | 20
Participants
  Treatment Emergent Adverse Events (TAEs) | 82 | 54 | 36 | 20
  Treatment Emergent Serious Adverse Events (TESAEs) | 37 | 38 | 24 | 9
  Deaths due to AE causally related to treatment | 2 | 0 | 0 | 0

6. Secondary Outcome: Apparent Clearance (CL/F) of Dabrafenib
Description: Blood samples from participants were collected for population pharmacokinetic analysis including the apparent base clearance (CL/F) following oral dosing of dabrafenib. Concentrations of dabrafenib was determined in plasma samples using the currently approved analytical methodology.
Time Frame: Week 3, Week 6, Week 12 and Week 18
Population: All subjects who received at least one dose of dabrafenib in the Cohort A (Dabrafenib Monotherapy) and in the doublets combination (Dabrafenib + Trametinib) Cohort B and C and provided an evaluable PK profile.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour (L/hr)
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 76 | 53 | 30
Liter/hour (L/hr) | 30.5 [29.1 to 32.0] | 21.4 [19.37 to 23.70] | 23.9 [22.02 to 25.87]

7. Secondary Outcome: Oral Volume of Distribution (V/F) of Dabrafenib
Description: Blood samples from participants were collected for population pharmacokinetic analysis including the oral volume of distribution (V/F) following oral dosing of dabrafenib. Blood samples from participants were collected for population pharmacokinetic analysis including the apparent base clearance (CL/F) following oral dosing of dabrafenib. Concentrations of dabrafenib was determined in plasma samples using the currently approved analytical methodology.
Time Frame: Week 3, Week 6, Week 12 and Week 18
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Liter (L)
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 76 | 53 | 30
Liter (L) | 50.6 [47.4 to 54.0] | 38.1 [30.93 to 46.97] | 48.1 [42.15 to 54.95]

8. Secondary Outcome: Apparent Clearance (CL/F) of Trametinib
Description: Blood samples from participants were collected for population pharmacokinetic analysis including the apparent base clearance (CL/F) following oral dosing of trametinib. Blood samples from participants were collected for population pharmacokinetic analysis including the apparent base clearance (CL/F) following oral dosing of dabrafenib. Concentrations of trametinib was determined in plasma samples using the currently approved analytical methodology.
Time Frame: Week 3, Week 6, Week 12 and Week 18
Population: All subjects who received at least one dose of trametinib in the doublets combination (Dabrafenib + Trametinib) Cohort B and C and provided an evaluable PK profile.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour (L/hr)
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 0 | 54 | 30
Liter/hour (L/hr) |  | 4.9 [4.62 to 5.19] | 5.03 [4.64 to 5.46]

9. Secondary Outcome: Oral Volume of Distribution (V/F) of Trametinib
Description: Blood samples from participants were collected for population pharmacokinetic analysis including the oral volume of distribution (V/F) following oral dosing of trametinib. Concentrations of trametinib was determined in plasma samples using the currently approved analytical methodology.
Time Frame: Week 3, Week 6, Week 12 and Week 18
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Liter (L)
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 0 | 54 | 30
Liter (L) |  | 91.98 [78.58 to 107.66] | 103.48 [84.58 to 126.59]

10. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration with dabrafenib and trametinib of 81 months (study treatment with dabrafenib and trametinib ranged from 0.3 to 80.0 months).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 9 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 81 months (study treatment with dabrafenib and trametinib), up to approximately 9 years (study duration)
Population: Clinical database population; all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Dabrafenib Monotherapy) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
Number analyzed (Participants) | 84 | 57 | 36 | 20
Participants
  On-treatment deaths | 15 | 12 | 5 | 4
  Post-treatment deaths | 38 | 38 | 21 | 13
  All deaths | 53 | 50 | 26 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days, up to approximately 81 months (study treatment with dabrafenib and trametinib ranged from 0.3 to 80.0 months).
Description: Any sign or symptom that occurs during the treatment period plus 30 days post-treatment.
Arm/Group | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD
All-Cause Mortality (participants affected / at risk) | 15/84 | 12/57 | 5/36 | 4/20
Serious Adverse Events (participants affected / at risk) | 37/84 | 38/57 | 24/36 | 9/20
Other Adverse Events (participants affected / at risk) | 82/84 | 54/57 | 36/36 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID (N=84) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD (N=57) | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD (N=36) | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Splenic thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1
Retinal dystrophy (Eye disorders) | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic duct stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Asthenia (General disorders) | 1 | 2 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 2 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 10 | 4 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Legionella infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 1
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 2 | 4 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal artery thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 3 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Dabrafenib Monotherapy): Dabrafenib Monotherapy 150mg BID (N=84) | Cohort B - Double Combination (Dabrafenib+Trametinib) mBRAF V600E: DAB 150MG BID, TRA 2mG QD (N=57) | Cohort C - Double Combination (Dabrafenib+Trametinib) Naive mBRAF V600E: DAB 150MG BID, TRA 2mG QD (N=36) | Crossover - Double Combination (Dabrafenib+Trametinib): DAB 150MG BID, TRA 2mG QD (N=20)
Anaemia (Blood and lymphatic system disorders) | 11 | 8 | 7 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 5 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 6 | 2 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 11 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 5 | 1 | 3
Cataract (Eye disorders) | 2 | 2 | 1 | 2
Dry eye (Eye disorders) | 4 | 6 | 3 | 0
Eye pain (Eye disorders) | 1 | 1 | 2 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 2 | 0
Photopsia (Eye disorders) | 0 | 1 | 2 | 0
Vision blurred (Eye disorders) | 5 | 2 | 3 | 0
Visual acuity reduced (Eye disorders) | 3 | 5 | 0 | 0
Visual impairment (Eye disorders) | 3 | 4 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 6 | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 8 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 10 | 11 | 6 | 6
Diarrhoea (Gastrointestinal disorders) | 17 | 18 | 15 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 3 | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 24 | 24 | 21 | 9
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 18 | 24 | 11 | 6
Asthenia (General disorders) | 25 | 21 | 4 | 3
Chest pain (General disorders) | 4 | 5 | 0 | 1
Chills (General disorders) | 12 | 15 | 10 | 3
Fatigue (General disorders) | 24 | 11 | 15 | 2
Feeling cold (General disorders) | 1 | 0 | 2 | 0
Gait disturbance (General disorders) | 1 | 0 | 2 | 1
Hyperthermia (General disorders) | 0 | 3 | 1 | 0
Influenza like illness (General disorders) | 2 | 4 | 5 | 0
Malaise (General disorders) | 5 | 3 | 4 | 1
Mucosal inflammation (General disorders) | 6 | 6 | 2 | 1
Non-cardiac chest pain (General disorders) | 5 | 0 | 1 | 1
Oedema peripheral (General disorders) | 3 | 22 | 13 | 5
Pain (General disorders) | 2 | 0 | 4 | 1
Pyrexia (General disorders) | 31 | 25 | 22 | 9
Bronchitis (Infections and infestations) | 6 | 6 | 0 | 3
Conjunctivitis (Infections and infestations) | 2 | 3 | 1 | 1
Folliculitis (Infections and infestations) | 4 | 4 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 2 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 8 | 7 | 7 | 3
Pneumonia (Infections and infestations) | 2 | 6 | 5 | 0
Rhinitis (Infections and infestations) | 5 | 7 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 5 | 7 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 5 | 2 | 0
Amylase increased (Investigations) | 0 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 6 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 5 | 11 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 6 | 1 | 2
Blood creatinine increased (Investigations) | 3 | 6 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 2 | 0
Lipase increased (Investigations) | 2 | 4 | 0 | 1
Weight decreased (Investigations) | 15 | 9 | 9 | 2
Weight increased (Investigations) | 0 | 8 | 3 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 25 | 17 | 12 | 6
Dehydration (Metabolism and nutrition disorders) | 5 | 3 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4 | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 9 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 5 | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 17 | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6 | 9 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 7 | 5 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 6 | 4 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 2 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 1 | 2 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 8 | 7 | 9 | 1
Dysgeusia (Nervous system disorders) | 3 | 5 | 0 | 0
Headache (Nervous system disorders) | 17 | 11 | 8 | 3
Memory impairment (Nervous system disorders) | 2 | 2 | 1 | 2
Paraesthesia (Nervous system disorders) | 4 | 3 | 2 | 0
Sciatica (Nervous system disorders) | 0 | 3 | 1 | 2
Taste disorder (Nervous system disorders) | 1 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 1 | 3
Confusional state (Psychiatric disorders) | 2 | 4 | 1 | 1
Depression (Psychiatric disorders) | 3 | 3 | 2 | 2
Insomnia (Psychiatric disorders) | 7 | 4 | 5 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 18 | 10 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 15 | 9 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 11 | 2 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 6 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 26 | 22 | 14 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 7 | 5 | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 7 | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 26 | 7 | 1 | 2
Madarosis (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 20 | 2 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 11 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 9 | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 15 | 16 | 11 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 1 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 0
Haematoma (Vascular disorders) | 1 | 1 | 2 | 1
Hypertension (Vascular disorders) | 4 | 6 | 4 | 4
Hypotension (Vascular disorders) | 6 | 6 | 5 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.